CLINICAL TRIAL: NCT06636240
Title: Study on the Potential Prebiotic Effects and Gut Microbiota Changes of Glucoside-enriched Mulberry Fruit in Children and Adolescents With Atopic Dermatitis
Brief Title: Prebiotic Effects of Mulberry Fruit in Children and Adolescents With Atopic Dermatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Meng-Che Lu, Pediatric Immunologist, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 113TMU-SHH-29
Record Dates: First submitted 2024-09-10; First posted 2024-10-10 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis (Eczema); Atopic Dermatitis, Probiotics
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control arm (Active Comparator): standard atopic dermatitis treatment
  Interventions: Other: Mometasone furoate 0.1% cream
- experimental arm (Experimental): add-on 200 ml/day mulberry juice with standard therapy
  Interventions: Dietary Supplement: Mulberry fruit juice

INTERVENTIONS:
Dietary Supplement: Mulberry fruit juice — Mulberry fruit juice 200ml/day plus standard therapy for atopic dermatitis including topical Mometasone furoate cream 0.1%
  Arms: experimental arm
Other: Mometasone furoate 0.1% cream — Standard therapy for atopic dermatitis including Mometasone furoate cream 0.1%
  Arms: control arm

SUMMARY:
This project proposes a randomized controlled human study to explore the prebiotic effects of consuming mulberry juice on atopic dermatitis in children and adolescents. The study aims to investigate the potential of mulberry fruit as a human prebiotic. This human study will recruit up to 120 participants from the Taipei Medical University Hospital (commissioned by the Ministry of Health and Welfare). Participants will be divided into experimental groups and a control group, with a 3-month intervention involving five clinical assessments and three stool collections. The goal is to compare the severity of atopic dermatitis, gut microbiota, and metabolite changes during the 6 days of mulberry juice consumption between the experimental and control groups.

This project will help establish mulberry fruit as a potential human prebiotic and adjunctive treatment for alleviating atopic dermatitis in children.

DETAILED DESCRIPTION:
The results of animal experiments have confirmed that mulberry fruit can improve atopic dermatitis. Its anti-inflammatory response is associated with the regulation of innate immune pathways and the restoration of skin barrier function. Additionally, mulberry extract may have prebiotic effects, altering the gut microbiota and metabolites to improve host health. Currently, mulberries are known to contain a significant amount of glucosides, with interleukin-17 isomer modulation being a major component. Therefore, mulberry fruit may have immune-regulatory effects, especially in Asian children and adolescents with elevated Th-17-related interleukin expression. However, it is paucity in research on the anti-inflammatory effects of mulberry fruit and its impact on gut microbiota in human atopic dermatitis.

This project proposes a randomized controlled human study to explore the long-term effects of consuming mulberry juice on atopic dermatitis in children and adolescents, as well as the composition of gut microbiota and metabolites. The study aims to investigate the potential of mulberry fruit as a human prebiotic. A randomized controlled human study will recruit up to 120 participants from the Taipei Medical University Hospital (commissioned by the Ministry of Health and Welfare). Participants will be divided into experimental groups and a control group, with a 3-month intervention involving five clinical assessments and three stool collections. The goal is to compare the severity of atopic dermatitis, gut microbiota, and metabolite changes during the 3 months of mulberry juice consumption between the experimental and control groups.

This project will help establish mulberry fruit as a potential human prebiotic and adjunctive treatment for alleviating atopic dermatitis in children. It will also lay the foundation for future research on effective component isolation and analysis, elucidating the impact of mulberry fruit on the composition of the human gut microbiota and metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 years and above (including 6 years) to less than 18 years (excluding 18 years)
* The legal guardian has the ability to understand and is willing to sign the written informed consent document
* Diagnosed by a physician according to the international Hanifin & Rajka criteria for atopic dermatitis, with a confirmed diagnosis of more than six months

Exclusion Criteria:

* Allergic to berries, mulberries, fruits from the same family (such as figs), or similar chemical or biological components
* Patients with immunodeficiency, including congenital or acquired immune disorders
* Patients with immune-related diseases other than allergies, asthma, or allergic rhinitis, including malignancies, rheumatic diseases, lupus erythematosus, chronic liver diseases, cirrhosis, kidney diseases, diabetes, or asplenia
* Individuals with other diseases or mental disorders that prevent them from complying with the intervention plan
* Patients with Short Bowel Syndrome
* Received oral or injectable antibiotics in the past month
* Received immunomodulators, biologics, or oral/injectable steroids exceeding 2 mg/kg/day in the past three months
* Underwent major surgery within 28 days before the study intervention (including the 28th day) or have not recovered from the side effects or complications of drug treatment/surgery from four weeks prior
* Currently participating in other drug intervention studies
* Currently experiencing systemic infection or unexplained fever (ear temperature greater than or equal to 38°C)
* Pregnancy
* Premature infants (born before 37 weeks, excluding 37 weeks)
* Individuals with congenital diseases, nutritional or metabolic disorders, or keratinization disorders
* Diagnosed with malignancies within the past five years.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change of Metabolism | 6 days until completion of juice intake
  Stool abundance statistical analysis at genus and species level, including richness, Chao1 index, Shannon and Simpson index, of gut microbiota from stool specimen collected from participants on 1st day and 8th day.

SECONDARY OUTCOMES:
Change of the Scoring Atopic Dermatitis (SCORAD) | From enrollment to the end of experiment at 12 weeks
  Evaluate the Scoring Atopic Dermatitis (SCORAD) scores on 1st day, 3rd, 6th, 9th and 12th week. The Score range is between 0 and 103 points and defines three classes of AD severity (i.e. mild if SCORAD <25, moderate if 25 ≤ SCORAD ≤ 50 and severe if SCORAD > 50)
Change of the Children's Dermatology Life Quality Index (CDLQI) | From enrollment to the end of experiment at 12 weeks
  Evaluate the Children's Dermatology Life Quality Index (CDLQI) scores on 1st day, 3rd, 6th, 9th and 12th week. The minimum score is 0 and the maximum score is 30. Higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Taipei Medical University Shuang Ho Hospital, Principal Investigator — Taipei Medical University
Locations (2):
- Taiwan (2):
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City, Taiwan
  - Taipei Medical University Shuang Ho Hospital, New Taipei City

IPD SHARING:
Plan to Share IPD: No